CLINICAL TRIAL: NCT02645071
Title: FAMILY Project: Brief Program in Reducing Sedentary Behavior and Promoting Physical Exercise
Brief Title: Brief Program in Reducing Sedentary Behavior and Promoting Physical Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: The Hong Kong Jockey Club Charities Trust (Other)
Responsible Party: Principal Investigator, Dr. Agnes Yuen-Kwan Lai, Research Officer, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UW15-743
Record Dates: First submitted 2015-12-29; First posted 2016-01-01 (Estimated); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: Physical Activity
Keywords: physical activity; family well being,; health
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Physical activity (Experimental): The experimental arm is a 15-20 min interactive session, which aims to reduce participants' sedentary behavior and increase physical activity by increasing their motivation, self-efficacy, and knowledge of different types of easy exercises.
  Interventions: Behavioral: Physical Activity

INTERVENTIONS:
Behavioral: Physical Activity — A brief education program in reducing sedentary behavior and promoting physical exercise with family would be conducted. Assessments will be conducted in two different time points, before training session (T1), immediately following training (T2) and two weeks after training (T3) to evaluate the effectiveness of training program.

SUMMARY:
Lack of physical activity was found to be a local and worldwide issue. Most Hong Kong people are having sedentary lifestyle. Researchers show that the increase of physical activity reduces the risk of chronic diseases, and improve cardio-pulmonary functions; whereas sedentary behaviors increase the risks.

For many people, the targets of the WHO physical activity guidelines are too high to be achieved. Some people are not even willing to try, despite the evidence for the protective benefits to their long term health. In response, a recent focus has been placed upon reduction of sedentary behavior. Sedentary behavior is defined as 'those activities that do not increase energy expenditure substantially above the resting level, such as sitting, lying down, or viewing TV, or simply as "too much sitting". The primary determinants of sedentary behavior are behavioral and context-based, such as TV and screen-focused behaviors in home and work environments, sitting at work, and sitting during transport. The public health leaders have called for reducing the time spent in sedentary behaviors as a possible public health priority. This study will focus on reduction of sedentary behavior and increasing physical activity in daily life. We hypothesize that the training programs would promote the health awareness of the participants.

DETAILED DESCRIPTION:
Physical activity is believed to contribute to physical and mental health, as well as social well-being. World Health organization (WHO) proposed that tobacco use, alcohol abuse, poor diets and physical inactivity are the common risk factors for non-communicable diseases (NCD) (WHO, 2014). The health benefits of regular physical activity (PA) are well established, including positive associations with psychological well-being and an inverse relationship with various illnesses.

Lack of physical activity was found to be a local and worldwide issue and most Hong Kong people are having a sedentary lifestyle. Studies show that the increase of physical activity reduces the risk of chronic diseases, and improve cardio-pulmonary functions; whereas sedentary behaviors increase the risks. In response, a recent focus has been placed upon reduction of sedentary behavior. The primary determinants of sedentary behavior are behavioral and context-based, such as TV and screen-focused behaviors in home and work environments, sitting at work, and sitting during transport. As a result, public health leaders have called for reducing the time spent in sedentary behaviors as a possible public health priority.

This study will focus on reduction of sedentary behavior and increasing physical activity in daily life. The intervention will promote activities that can be done without using extra time (Zero-time exercise). These exercises will encourage participants to use larger muscle groups than they would simply sitting or standing, but are designed to be done by all ages and all fitness levels. For example, while standing, participants will be encouraged to balance on one leg, which will engage stomach and leg muscles. There is evidence that these types of movements create cardiovascular and skeletal muscle changes.

The intervention is a 15- to 20- minute interactive session program, which aims to reduce participants' sedentary behavior and increase physical activity by increasing their motivation, self-efficacy and knowledge of different types of easy movements (Zero-time exercises). We hypothesize that the training programs would promote the health awareness of the participants.

The primary objective is to promote the health awareness on reducing sedentary behavior and/or increasing physical exercise. The secondary objectives are to enhance intention and confidence of participants to encourage their family members to reduce sedentary and/or increasing physical exercise.

ELIGIBILITY:
Inclusion Criteria:

* Chinese speaking
* Able to complete the questionnaire
* Aged 18 or above

Exclusion Criteria:

- People with serious health condition that might prevent them from participating in physical activity

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Change in intention on performing physical activity in relation to reduce sedentary behavior | baseline, immediately following the training session, 2 weeks
  Intention on performing physical activity in relation to reduce sedentary behavior, will be assessed by outcome-based physical activity questionnaire

SECONDARY OUTCOMES:
Change in confidence on performing physical activity in relation to reduce sedentary behavior | baseline, immediately following training, 2 weeks
  Confidence on performing physical activity in relation to reduce sedentary behavior, will be assessed by outcome-based physical activity questionnaire
Change in perceived knowledge on performing physical activity in relation to reduce sedentary behavior | baseline, immediately following training, 2 weeks
  Perceived knowledge on performing physical activity in relation to reduce sedentary behavior, will be assessed by outcome-based physical activity questionnaire
Change in behaviour on performing physical activity in relation to reduce sedentary behavior | baseline, 2 weeks
  Behaviour on performing physical activity in relation to reduce sedentary behavior, will be assessed by outcome-based physical activity questionnaire
Change in participants' own health and happiness | baseline, 2 weeks
  Personal health and happiness will be assessed by personal health and happiness scale
Change in participants' family well-being | baseline, 2 weeks
  Family well-being will be assessed by family well-being scale
Change in intention to motivate participants' family members to reduce sedatry behvaiour | baseline, immediately following training, 2 weeks
  Intention to motivate participants' family members on reducing sedentary behaviour, will be assessed by outcome-based physical activity questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Agnes YK LAI, DN, Principal Investigator — The University of Hong Kong
Locations (1):
- Department of Health, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bellicha A, Kieusseian A, Fontvieille AM, Tataranni A, Charreire H, Oppert JM. Stair-use interventions in worksites and public settings - a systematic review of effectiveness and external validity. Prev Med. 2015 Jan;70:3-13. doi: 10.1016/j.ypmed.2014.11.001. Epub 2014 Nov 10. PMID 25449692
- [Background] Gardiner PA, Eakin EG, Healy GN, Owen N. Feasibility of reducing older adults' sedentary time. Am J Prev Med. 2011 Aug;41(2):174-7. doi: 10.1016/j.amepre.2011.03.020. PMID 21767725
- [Background] Kamani CH, Gencer B, Montecucco F, Courvoisier D, Vuilleumier N, Meyer P, Mach F. Stairs instead of elevators at the workplace decreases PCSK9 levels in a healthy population. Eur J Clin Invest. 2015 Oct;45(10):1017-24. doi: 10.1111/eci.12480. Epub 2015 Aug 26. PMID 26081791
- [Background] Torbeyns T, Bailey S, Bos I, Meeusen R. Active workstations to fight sedentary behaviour. Sports Med. 2014 Sep;44(9):1261-73. doi: 10.1007/s40279-014-0202-x. PMID 24842828
- See also: World Health Organization (2015). Physical activity : Fact sheet — http://www.who.int/mediacentre/factsheets/fs385/en/
- See also: Department of Health (2014). Behavioral Risk Factor Survey — http://www.chp.gov.hk/en/behavioural/10/280.html